CLINICAL TRIAL: NCT06994923
Title: Testing a Behavioral Weight Loss Intervention for Emerging Adults Implemented Within College Health Service Centers
Brief Title: Weight Management Intervention in College: A Pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17937323; K23DK128561 (NIH)
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-05

CONDITIONS: Obesity and Overweight
Keywords: obesity; college students; behavioral weight loss intervention; small changes
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: A 2-arm parallel randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BWLI-College (Experimental): BWLI-College is a multicomponent behavioral weight loss intervention to reduce weight through diet, physical activity, and behavioral modifications designed to be responsive to emerging adult preferences. It will be delivered in a hybrid format with in-person and remotely-delivered synchronous sessions. As presently designed, the intervention will last 10 weeks.
  Interventions: Behavioral: BWLI-College
- Control (Active Comparator): The Control intervention consists of 1 in-person psychoeducational group session on general weight loss information and myths. Public web-resources about healthy eating and physical activity will be provided. Newsletters with similar content will be sent to promote retention.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: BWLI-College — Behavioral modifications are based on empirically-supported principles for weight loss. Diet recommendations follow a small change approach in which participants will make a series of small, self-selected dietary changes each day (~100-200 calories) that they build on over the course of the intervention. Physical activity recommendations are to achieve 150-250 weekly minutes of moderate-to-vigorous physical activity with specific goals and rate of progression that are individualized to each participant.
  Arms: BWLI-College
Behavioral: Control — Psychoeducation around dieting myths, healthy eating, and physical activity
  Arms: Control

SUMMARY:
This pilot randomized controlled trial will examine a behavioral weight loss intervention that uses a "small change" approach fro emerging adult college students with overweight/obesity. The primary aim is to assess student acceptability and clinically-meaningful weight changes.

DETAILED DESCRIPTION:
Forty percent of emerging adults (age 18-25) have overweight or obesity, which is unlikely to remit and has significant health consequences. However, emerging adults are underrepresented in traditional weight loss programs, drop-out at high rates, and have blunted weight loss outcomes. One potential way to improve participation is to offer BWLIs in college health service centers to reduce barriers to participation. Approximately 40% of emerging adults are enrolled in a postsecondary institution and college health centers are used widely by students. Moreover, delivering an intervention with design features that are responsive to emerging adult preferences and lifestyles may also improve intervention effectiveness and attractiveness. The "small change" (SC) approach to weight loss addresses emerging adult barriers to engagement by focusing on reducing calories through a few self-selected, specific changes to current obesogenic behaviors, requiring less time and effort than traditional behavioral weight loss interventions (BWLI) and promoting autonomy and self-efficacy. The SC approach has been used effectively for weight loss in other populations. This randomized controlled pilot study is part of a larger study that aims to develop and refine a novel and effective BWLI based on a SC approach that is designed for emerging adults and for implementation in college health centers, an accessible care setting. The primary aim of this substudy is to assess acceptability and feasibility of the intervention and to get a preliminary understanding of potential clinical benefit for participants.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 25 or greater
* Enrolled at college/university where study will take place
* English-speaking

Exclusion Criteria:

* History or current diagnosis of anorexia nervosa, bulimia nervosa, or alcohol use disorder (current symptoms also assessed at screening using validated screening questionnaires)
* Participation in another formal weight loss program or current utilization of obesity medications
* Current or recent pregnancy
* Psychiatric hospitalization in the past 12 months
* Recent weight loss of 5% body weight or more
* History of bariatric surgery
* Severe food or physical activity restrictions that would interfere with treatment recommendations

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability | 10 weeks
  Refers to the satisfactory nature of a treatment and will be assessed via the 4-item Acceptability of Intervention Measure. Benchmarks are to reach mean scores of at least 4 out of 5.
Retention | 10 weeks
  Rate of retention of 70% or more (benchmark)
Adherence | 10 weeks
  Average attendance of 75% or more (benchmark)
Weight Loss | 10 weeks
  Average weight loss of at least 3%

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline F Hayes, PhD, Principal Investigator — Brown University
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided